CLINICAL TRIAL: NCT04834427
Title: Safety and Efficacy Evaluation of S (+) -Ketamine for Postoperative Acute Pain in Children in Perioperative Settings: A Multicenter, Randomized, Open-label, Active Controlled Pragmatic Clinical Trial
Brief Title: Safety and Efficacy Evaluation of S (+) - Ketamine in Children
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Southern Medical University, China (Other); Beijing Children's Hospital (Other); Shanghai Children's Medical Center (Other); Hunan Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Weidong Mi, Director of the Department of Anesthesiology, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-SK-C
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: S-ketamine; Esketamine; Acute Pain; Postoperative Pain; Analgesia; Hyperalgesia; Delirium; Depression, Anxiety; Children
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Agnosia; Hyperalgesia; Delirium; Depression; Anxiety Disorders | interventions — Ketamine; Esketamine

STUDY DESIGN:
Intervention Model Description: Experimental group : Control group=2:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S (+)-Ketamine group (Experimental): Patients who undergo general anesthesia using S(+)-ketamine hydrochloride for anesthesia induction, maintenance or postoperative analgesia.
  Interventions: Drug: Conventional therapy + S (+)-Ketamine
- Control group (Active Comparator): Patients who undergo conventional therapy without S (+)-Ketamine hydrochloride injection during perioperative period.
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Drug: Conventional therapy + S (+)-Ketamine — In principle, there are no specific restrictions on the dosage, mode of administration, timing, and compatibility of S-ketamine hydrochloride injection, but the recommended dosage is given, which is lower than the dosage specified in the instructions.
  Recommended use and dosage of S (+)-Ketamine:
  1. Intravenous injection：Bolus intravenous injection before skin incision, the dose is 0.1~0.25 mg/kg; Bolus intravenous injection (dose 0.1~0.25 mg/kg) before skin incision + continuous intravenous infusion (dose of 0.1~0.25 mg/kg/h) during operation; Continuous intravenous infusion after surgery with a dose of 0.02~0.1 mg/kg/h for 24~48 h.
  2. Intramuscular injection：The dose is 2~4 mg/kg.
  Other Names: Conventional therapy + S-ketamine; Conventional therapy + Esketamine
  Arms: S (+)-Ketamine group
Drug: Conventional therapy — Receiving conventional therapy without S (+)-Ketamine hydrochloride injection. There is no restrictions in drugs, doses and incompatibility, the researchers can choose appropriate medication regimens based on clinical practice, but other NMDA receptor antagonists are not be allowed to use, such as dextromethorphan and amantadine.
  Other Names: Routine treatment
  Arms: Control group

SUMMARY:
A multicenter, randomized, open-label, active controlled pragmatic clinical trial that evaluates the safety and efficacy of S (+) -ketamine for postoperative acute pain in children in perioperative settings.

DETAILED DESCRIPTION:
Children often suffer acute pain,awakening delirium, anxiety and depression after operation which may affect the recovery of children. S (+) - ketamine has been described to decrease acute pain and opioid consumption,but it needs to confirm for chinese children undergoing surgery.

Objective:

To evaluate the analgesic effect of perioperative administration of S (+) - ketamine on postoperative acute pain in children undergoing surgery, and explore the effects of S (+) - ketamine on postoperative awakening delirium, postoperative anxiety and depression mood ,as well find the best usage, including dose, timing, compatibility, and type of operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤17 years;
2. Scheduled for elective digestive tract surgery, orthopedic surgery, urological surgery , ear surgery or other surgeries under general anesthesia;
3. ASA physical status I～Ⅲ;
4. The informed consent form was signed by the patients or the guardians.

Exclusion Criteria:

1. The expected length of hospital stay of the patient is less than 48h;
2. Patients expected to be admitted to the ICU after surgery;
3. Patients expected to return to the ward with tracheal catheter after surgery;
4. Be allergic to S (+) - ketamine;
5. Patients with severe disorder of consciousness or mental system diseases (schizophrenia, mania, bipolar disorder, psychosis, etc.) or cognitive dysfunction;
6. Patients with congenital heart disease or severely developmental retardation;
7. Patients with any of the following contraindications of S (+) - ketamine:

   1. Patients with risk of serious rise of blood pressure or intracranial pressure;
   2. Patients with high intraocular pressure (glaucoma) or penetrating ocular trauma;
   3. Patients with poorly controlled or untreated hypertension (Resting systolic blood pressure greater than 180 mmHg, or resting diastolic blood pressure greater than 100mmHg);
   4. Patients with untreated or undertreated hyperthyroidism.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
The area under the broken line of FLACC scale score | Hour 0-48 after surgery
  Only for children aged 0~7 years. The score of FLACC Scale is 0-10, the higher the score, the more severe the pain.
The area under the broken line of Numerical Rating Scale score | Hour 0-48 after surgery
  Only for children aged 8~17years. The score of Numerical Rating Scale(NRS) is 0-10, the higher the score, the more severe the pain.
Opioid consumption | Hour 0-48 after surgery
  Total opioid consumption(conversion to equivalent morphine)

OTHER OUTCOMES:
FLACC scale score | Hour 0-48 after surgery
  Only for children aged 0~7 years. The score of FLACC Scale is 0-10, the higher the score, the more severe the pain.
  8≤Age ≤17 years: NRS pain score at 2h, 4h, 24h, 48h after surgery.
Numerical Rating Scale score | Hour 0-48 after surgery
  Only for children aged 8~17years. The score of Numerical Rating Scale(NRS) is 0-10, the higher the score, the more severe the pain.
Time of first rescue analgesia | Hour 0-48 after surgery
  The time from the end of the operation to the first rescue analgesics after the operation. Rescue analgesia refers to the analgesia according to the patient's or guardian's requirements in addition to routine postoperative analgesia.
The incidence of rescue analgesia | Hour 0-48 after surgery
  Rescue analgesia refers to the analgesia according to the patient's or guardian's requirements in addition to routine postoperative analgesia.
Recovery time | Day 0
  The time from the end of the operation to recovery(can be awakened)
The incidence of emergence delirium | Day 0
  Only for children aged 0-7 years. Evaluating by the Pediatric Emergence Delirium Rating Scale(PAED) ,the score of the scale is 0~20, when the total score is greater than 10, it is considered that the child has delirium.The scale will be evaluated 10minutes, 20minutes, 30minutes after extubation.
The incidence of unexpected intraoperative events | Intraoperative
  Unexpected events during operation include intraoperative cough, laryngeal spasm, body movement, tachycardia, decreased oxygen saturation, respiratory depression, bradycardia, hypertension and hypotension.
The incidence of adverse events after surgery | Hour 0-48 after surgery
  The incidence of adverse events from the end of the operation to 48h after surgery. Including nausea, vomiting, increased secretions, dizziness, oversedation, infection,anesthetic awareness, nightmares, restlessness, pruritus, disorientation, delirium, respiratory depression, diplopia, diarrhea, intestinal obstruction, urinary retention, gastroesophageal reflux, constipation, chills, hallucinations, etc.
Children's Depression Inventory(CDI) score | Hour 48 after surgery
  Only for children aged 8~17.Children's Depression Inventory(CDI) scale include 27 questions ,from 0 to 54pionts, the higher the score, the more severe the depressive symptoms.
Hospital Anxiety and Depression Scale(HAD）score | Hour 48 after surgery
  Only for children aged 14~17.Hospital Anxiety and Depression Scale(HAD）include anxiety measure(7 questions,0-21pionts) and depression measure(7 questions,0-21pionts),the higher the score, the more severe the symptoms.
Pharmacoeconomic indicators | Hour 48 after surgery
  Calculating incremental cost-effectiveness ratio （ICER）based on cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Duan C, Zhang J, Qu S, Sun Y, Zhou L, Yang L, Lan C, Mi W, Chen P. Evaluation of the effect of perioperative administration of S(+)-ketamine hydrochloride injection for postoperative acute pain in children: study protocol for a prospective, multicenter, randomized, open-label, parallel-group, pragmatic clinical trial. Trials. 2022 Jul 23;23(1):586. doi: 10.1186/s13063-022-06534-z. PMID 35870990